CLINICAL TRIAL: NCT02703805
Title: Fit For Function: A Community Wellness Program for Persons With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); YMCA of Hamilton/Burlington/Brant (Unknown); YMCA of Niagara (Unknown); Brant Community Healthcare System (Unknown); Niagara Health System (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FFF133486
Record Dates: First submitted 2014-10-14; First posted 2016-03-09 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Cerebrovascular Accident
Keywords: Community program; Wellness; Exercise; Physical Activity; Education; Stroke; Self-management
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fit For Function Program (Experimental): A 12-week YMCA-based wellness program for persons with stroke, consisting of 2 group exercise sessions, one gym exercise session and one education session per week with trained instructors.
  Interventions: Other: Fit For Function Program
- Standard YMCA membership (Active Comparator): A 12 week standard YMCA membership.
  Interventions: Other: Standard YMCA membership

INTERVENTIONS:
Other: Fit For Function Program — A 12-week YMCA-based wellness program for persons with stroke, consisting of 2 group exercise sessions, one gym exercise session and one education session per week with trained instructors
  Arms: Fit For Function Program
Other: Standard YMCA membership — A 12 week standard YMCA membership.
  Arms: Standard YMCA membership

SUMMARY:
Building on an earlier pilot study, this randomized controlled trial will compare the effectiveness of a 12 week community YMCA-based wellness program specifically designed for people with stroke (Fit for Function) to a standard YMCA membership.

DETAILED DESCRIPTION:
The program will be delivered through a partnership between McMaster University, the YMCA and Hamilton Health Sciences/ the Brant Community Healthcare System/ the Niagara Health System. Participants will exercise three times a week and receive weekly education about how to take care of themselves after a stroke. The YMCA staff who deliver the program will have specialized training about how to help people with a stroke exercise safely and effectively. The hospital within each region will provide specialized on-site physiotherapy consultative support. The comparator standard YMCA membership will include typical sessions with a wellness coach who has basic safety training regarding stroke and exercise.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stroke
* 18 years of age or older
* community dwelling
* able to walk 10m independently, with or without an assistive device
* medically approved by a physician to participate
* able to tolerate 60 minutes of activity with rest intervals
* able to independently follow instructions

Exclusion Criteria:

* involved in an active rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in the Reintegration to Normal Living Index (RNL) from baseline | baseline, 12 weeks, 24 weeks
  This measure assesses the degree to which individuals who have experienced traumatic or incapacitating illness achieve reintegration into normal social activities.

SECONDARY OUTCOMES:
Change in The Rapid Assessment of Physical Activity (RAPA) score from baseline | baseline, 12 weeks, 24 weeks
  This is a 9-item measure that assesses frequency and intensity of aerobic physical activity and frequency of strengthening and flexibility exercises.
Change in The Short Portable Performance Tests (SPPT) score from baseline | baseline, 12 weeks, 24 weeks
  This test is used to quantify lower extremity function by evaluating the time to walk 8 feet, standing balance and repeated chair stands.
Change in The Six Minute Walk Test (6MWT) from baseline | baseline, 12 weeks, 24 weeks
  This test is an indicator of exercise capacity and measures the distance walked in 6 minutes.
Change in Strength: Grip and Knee extension from baseline | baseline, 12 weeks, 24 weeks
  Hand-held dynamometry will measure the average strength of three trials.
Change in The EQ-5D score from baseline | baseline, 12 weeks, 24 weeks
  This is a generic utility-based health related quality of life questionnaire.
Change in The Patient Activation Measure (PAM) score from baseline | baseline, 12 weeks, 24 weeks
  This is a 13-item measure of the patient's level of knowledge, skill and confidence for self-management.
Change in The Body Mass Index (BMI) score from baseline | baseline, 12 weeks, 24 weeks
  The BMI will be calculated from measurements of body mass and height as an indicator of cardiovascular health.
Change in Blood lipid levels from baseline | baseline, 12 weeks, 24 weeks
  12 hour fasting levels of lipids will be used as an indicator of cardiovascular health.
Change in blood glucose levels from baseline | baseline, 12 weeks, 24 weeks
  12 hour fasting levels of glucose in blood will be used as an indicator of cardiovascular health.
Change in blood inflammatory markers from baseline | baseline, 12 weeks, 24 weeks
  12 hour fasting levels of inflammatory markers in blood will be used as an indicator of cardiovascular health.
Healthcare Utilization Questionnaire | 0- 24 weeks
  An indicator of healthcare resource utilization (hospitalizations, medical appointments and investigations, medication use) for economic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University; Ada Tang, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - The Brantford Family YMCA, Brantford, Ontario
  - Downtown Hamilton YMCA, Hamilton, Ontario
  - The Walker Family YMCA, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Results will be communicated to the Central South Regional Stroke Network and the Ontario Stroke System. Results will also be disseminated through professional organizations, the Ontario Ministry of Health and Long Term Care, peer reviewed conferences, provincial and national stroke forums, journal articles and special interest groups like the Stroke Recovery Group.

REFERENCES:
- [Derived] Richardson J, Tang A, Guyatt G, Thabane L, Xie F, Sahlas D, Hart R, Fleck R, Hladysh G, Macrae L. FIT for FUNCTION: study protocol for a randomized controlled trial. Trials. 2018 Jan 15;19(1):39. doi: 10.1186/s13063-017-2416-3. PMID 29335013